CLINICAL TRIAL: NCT00888732
Title: A Comparison of Pharmacodynamics and Pharmacokinetics of Insulin Aspart, Biphasic Insulin Aspart 70 and 50 & Fast-acting Human Insulin in Patients With Type 1 Diabetes, A Randomised, Quadruple Crossover Trial
Brief Title: A Comparison of Pharmacodynamics and Pharmacokinetics of Insulin Aspart, BIAsp70, BIAsp50 and Fast-acting Human Insulin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Jens Sandahl Christiansen, M.D., University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Asp-BIAsp-HI-2008; 2008-007176-22 (EudraCT Number)
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Insulin Aspart; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin therapy (Experimental): Insulin Aspart, Biphasic Insulin Aspart 70 and 50 & Fast-acting Human Insulin
  Interventions: Drug: Insulin Aspart, BIAsp 70, BIAsp50, Human Insulin

INTERVENTIONS:
Drug: Insulin Aspart, BIAsp 70, BIAsp50, Human Insulin — 0.2 U/IU/kg subcutaneous injection, single dose
  Other Names: - Insulin Aspart: NovoRapid; - BIAsp 50: NovoMix 50; - BIAsp 70: NovoMix 70; - Human Insulin: Actrapid

SUMMARY:
The hypothesis is that an optimal formulation of fast acting and intermediary acting insulin analogues will improve post prandial glycaemic control in patients with type 1 diabetes

DETAILED DESCRIPTION:
This trial is a single centre, open-label, randomised 4 period cross-over trial, comparing the pk and pd profiles of IAsp, BIAsp 50, BIAsp 70 and Fast-acting Human Insulin after a standard test meal in subjects with type 1 diabetes. The profiles will be derived over a 12-hour period after subcutaneous injection in the abdominal region with a single dose of IAsp, BIAsp 50, BIAsp 70 or Fast-acting Human Insulin at a test meal. The trial consists of a screening period of 4-21 days and 4 treatment visits.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities.
* Diagnosed type 1 diabetes before the age of 40 and on insulin treatment within one year of diagnosis.
* Insulin treatment of any regime for more than one year at time of inclusion.
* Total insulin demand ≥ 0,4 U/IU/kg/24 hrs
* HbA1c between 7% and 12% (both values included).
* Age ≥ 18 years.
* BMI between 18 and 35 kg /m2 (including both values).

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products.
* Recurrent major hypoglycaemic episodes.
* Heart: Unstable Angina Pectoris, AMI < 12 months or heart insufficiency classified according to NYHA III-IV
* Blood Pressure: Severe uncontrolled hypertension with BP > 180/110 mmHg, sitting
* Liver: Impaired hepatic function corresponding to serum-ALAT or basic phosphatase > 2 x upper reference limit of the local laboratory.
* Kidneys: Impaired renal function corresponding to serum-creatinin > 150 μmol/l according to the local laboratory.
* Any disease judged by the investigator to affect the trial.
* Pregnancy, breast-feeding or the intention of becoming pregnant or fertile women not using adequate contraceptive measures - adequate contraceptive method is sterilisation, hysterectomy or current use of contraceptive pills or intra uterine device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Cmaxglu: Peak plasma glucose following test meal (breakfast). A comparison will be made between fast-acting human insulin vs. IAsp, BIAsp 50 and BIAsp 70, IAsp vs BIAsp 50 and BIAsp 70, BIAsp 50 vs. BIAsp 70. | 12 hours following a standard test meal (breakfast)

SECONDARY OUTCOMES:
AUCglu: The area under the plasma glucose concentration (0-12, 0-6, 6-12, 0-4, 4-8, 8-12 hours after test meal) after a single injection of one of the four insulins: IAsp, Biphasic insulin aspart 50 and 70 & fast-acting human insulin | 12 hours following a standard test meal (breakfast)
AUCins: The area under insulin aspart/human insulin concentration (0-12, 0-6, 6-12, 0-4, 4-8, 8-12 hours after test meal) after a single injection of one of the four insulins: IAsp, Biphasic insulin aspart 50 and 70 & fast-acting human insulin | 12 hours following a standard test meal (breakfast)
tmaxins: Time to maximum serum insulin aspart/human insulin concentration | 12 hours following a standard test meal (breakfast)
Serum GH, total IGF-I, IGF-I bioactivity, IGFBP-1, IGFBP-2, binary complex of IGF-I, IGFBP-3 and the acid-labile subunit (ALS) | 12 hours following a standard test meal (breakfast)

CONTACTS AND LOCATIONS:
Overall Officials: Jens S Christiansen, M.D, Principal Investigator — University of Aarhus
Locations (1):
- Dept of Medicine M, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Background] Thorisdottir RL, Parkner T, Chen JW, Ejskjaer N, Christiansen JS. A comparison of pharmacokinetics and pharmacodynamics of biphasic insulin aspart 30, 50, 70 and pure insulin aspart: a randomized, quadruple crossover study. Basic Clin Pharmacol Toxicol. 2009 Mar;104(3):216-21. doi: 10.1111/j.1742-7843.2008.00355.x. Epub 2009 Jan 20. PMID 19175369
- [Background] Weyer C, Heise T, Heinemann L. Insulin aspart in a 30/70 premixed formulation. Pharmacodynamic properties of a rapid-acting insulin analog in stable mixture. Diabetes Care. 1997 Oct;20(10):1612-4. doi: 10.2337/diacare.20.10.1612. PMID 9314644
- [Background] Kang S, Creagh FM, Peters JR, Brange J, Volund A, Owens DR. Comparison of subcutaneous soluble human insulin and insulin analogues (AspB9, GluB27; AspB10; AspB28) on meal-related plasma glucose excursions in type I diabetic subjects. Diabetes Care. 1991 Jul;14(7):571-7. doi: 10.2337/diacare.14.7.571. PMID 1914797
- [Background] Thrailkill KM. Insulin-like growth factor-I in diabetes mellitus: its physiology, metabolic effects, and potential clinical utility. Diabetes Technol Ther. 2000 Spring;2(1):69-80. doi: 10.1089/152091599316775. PMID 11467325
- [Background] Jacobsen LV, Sogaard B, Riis A. Pharmacokinetics and pharmacodynamics of a premixed formulation of soluble and protamine-retarded insulin aspart. Eur J Clin Pharmacol. 2000 Aug;56(5):399-403. doi: 10.1007/s002280000159. PMID 11009049
- [Derived] Ma Z, Christiansen JS, Laursen T, Wu C, Lauritzen T, Parkner T, Frystyk J. Effects of human insulin and insulin aspart preparations on levels of IGF-I, IGFBPs and IGF bioactivity in patients with type 1 diabetes. BMC Endocr Disord. 2014 Apr 11;14:35. doi: 10.1186/1472-6823-14-35. PMID 24725803
- [Derived] Ma Z, Parkner T, Frystyk J, Laursen T, Lauritzen T, Christiansen JS. A comparison of pharmacokinetics and pharmacodynamics of insulin aspart, biphasic insulin aspart 70, biphasic insulin aspart 50, and human insulin: a randomized, quadruple crossover study. Diabetes Technol Ther. 2012 Jul;14(7):589-95. doi: 10.1089/dia.2011.0299. Epub 2012 Apr 20. PMID 22519735
- See also: Click here for more information about trial site (Danish version only) — http://www.aarhussygehus.dk